CLINICAL TRIAL: NCT04743674
Title: Plasma Circulating Tumor HPVDNA and Transrenal HPVDNA as Minimally Invasive Biomarkers for Cervical Cancer Detection and Surveillance Following Definitive Treatment
Brief Title: Blood and Urine HPVDNA as Minimally Invasive Biomarkers for Cervical Cancer Detection and Surveillance Following Treatment
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 2051
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, and archived/ left over biopsy tissue will be tested for HPVDNA and retained for up to 15 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine if ctHPVDNA (circulating tumor HPV DNA) can be used as a non-invasive biomarker for identification and treatment monitoring of cervical cancer by characterizing correlation between plasma ctHPVDNA, urine transrenal HPVDNA (TrHPVDNA) levels and presence of cervical cancer at diagnosis and following definitive intent management.

DETAILED DESCRIPTION:
Early stage cervical cancer is managed surgically while chemoradiation is the mainstay for treatment of bulky or advanced stage disease. The primary aim of post-treatment surveillance is to detect early recurrences and guide additional therapy. There is no definitive agreement on the best practice for cervical cancer surveillance. Most recurrences are detected based on patient history and physical exam as there is limited data to support cervicovaginal cytology and routine use of imaging in follow up. Novel non-invasive biomarkers are needed to monitor disease status, detect early recurrence and guide personalized treatment decisions. Biospecimens including urine and blood plasma will be collected from patients presenting to the UNC Department of Gynecology Oncology and Multidisciplinary clinics with newly diagnosed cervical cancer to assess for HPVDNA. Archived or residual tissue will also be accessed. For patients who undergo definitive management with surgery or chemoradiation, a post-treatment blood plasma and urine sample will be collected 2-6 weeks after completion and will be compared to pre-therapy ctHPVDNA and TrHPVDNA levels.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older on day of signing informed consent
* New diagnosis of cervical cancer
* Subject is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee

Exclusion Criteria:

* Women who are pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with newly diagnosed cervical cancer planning to be treated with surgery or chemoradiation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Relationship between ctHPVDNA levels in plasma, TrHPVDNA levels in urine, and presence of cervical cancer in women being evaluated in clinic. | Baseline
  We will quantify ctHPVDNA levels in blood plasma and TrHPVDNA in urine from patients with cervical cancer at time of diagnosis.

SECONDARY OUTCOMES:
Change in ctHPVDNA and TrHPVDNA levels following definitive intent therapy for early stage disease. | 2-6 weeks post-treatment
  We will collect bio-specimens and quantify ctHPVDNA and TrHPVDNA levels in plasma and urine, respectively, during their post-treatment visit typically 2-6 weeks post-surgery or last day of treatment visit (chemoradiation).

CONTACTS AND LOCATIONS:
Overall Officials: Shivani Sud, MD, Principal Investigator — UNC
Locations (2):
- Melissa Knutsen, Chapel Hill, North Carolina, United States
- Kamuzu Central Hospital, Lilongwe, Malawi

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials